CLINICAL TRIAL: NCT02186821
Title: Modular Phase II Study to Link Targeted Therapy to Patients With Pathway Activated Tumors: Module - 7 Ceritinib (LDK378) for Patients Whose Tumors Have Aberrations in ALK or ROS1
Brief Title: Ceritinib (LDK378) for Patients Whose Tumors Have Aberrations in ALK or ROS1 (SIGNATURE)
Acronym: SIGNATURE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated due to low enrollment
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLDK378AUS23
Record Dates: First submitted 2014-07-03; First posted 2014-07-10 (Estimated); Results first posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-03

CONDITIONS: Tumors With Aberrations in ALK or ROS1
Keywords: hematological malignancy; solid tumor malignancy; mutation; translocation; rearrangement; amplification; ALK; ROS1; NSCLC; B-cell lymphoma
MeSH Terms: conditions — Hematologic Neoplasms; Lymphoma, B-Cell | interventions — ceritinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ceritinib 750 mg (Experimental): Ceritinib was dosed on a flat scale of 750 mg (e.g., 5 x 150 mg capsules) orally, once daily, on a continuous dosing cycle. A complete treatment cycle was defined as 28 days with no breaks between dosing cycles.
  Interventions: Drug: Ceritinib

INTERVENTIONS:
Drug: Ceritinib — Ceritinib was dosed on a flat scale of 750 mg (e.g., 5 x 150 mg capsules) orally,once daily, on a continuous dosing cycle. A complete treatment cycle was defined as 28 days. There were no breaks between dosing cycles.
  Other Names: LDK378

SUMMARY:
The purpose of this signal seeking study was to determine whether treatment with ceritinib demonstrated sufficient efficacy in select pathway-activated solid tumors and/or hematologic malignancies to warrant further study.

DETAILED DESCRIPTION:
This was an open label study to determine the efficacy and safety of treatment with ceritinib in patients with a diagnosis of solid tumors or hematological malignancies that had been pre-identified (prior to study consent) to have ALK or ROS1 positive mutations, translocations, rearrangements or amplifications and whose disease had progressed on or after standard treatment. The study consisted of a treatment phase where all patients received ceritinib capsules for a total dose of 750 mg daily for up to 8 cycles of 28 days. Disease assessments for clinical benefit were performed every 8 weeks until disease progression or end of treatment. Following discontinuation of treatment for any reason, patients were followed for safety for 30 days. Survival information was collected every 3 months until 2 years after the last patient had enrolled into the study. Study was amended to allow for discontinuation of survival period if primary endpoint was not met.

Study was terminated due to low enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Patient had a confirmed diagnosis of a select solid tumor (except ALK+ NSCLC) or hematological malignancy and was in need of treatment because of radiologic progression or relapse.
* Patient must have been pre-identified as having a tumor with an ALK or ROS1 positive mutation, translocation, rearrangement or amplification. The qualifying alteration must have been assessed and reported by a CLIA-certified laboratory. ALK positivity as assessed by IHC or FISH were allowed.
* Patient must have received at least one prior treatment for recurrent, metastatic and/or locally advanced disease and for whom no standard therapy options were anticipated to result in a durable remission.
* Patient had progressive and measurable disease as per RECIST 1.1 or other appropriate hematological guidelines.
* Patient had an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1.

Exclusion Criteria:

* Patient had received prior treatment with ceritinib.
* Patients with symptomatic CNS metastases who were neurologically unstable or required increasing doses of steroids within the 2 weeks prior to study entry to manage CNS symptoms.
* Patient had received chemotherapy or anticancer therapy ≤ 4 weeks (6 weeks for nitrosourea, monoclonal antibodies or mitomycin-C) prior to starting study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2014-09-17 (Actual); Primary Completion 2017-12-13 (Actual); Study Completion 2017-12-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (21):
- United States (21):
  - St Joseph Heritage Healthcare St. Joseph Heritage, Santa Rosa, California
  - Sarah Cannon Research Institute, Denver, Colorado
  - Rocky Mountain Cancer Centers Dept of Rocky Mountain (2), Greenwood Village, Colorado
  - Florida Cancer Specialists Florida Cancer Specialists (31, Fort Myers, Florida
  - Northwestern University Northwestern (6), Chicago, Illinois
  - Physicians Clinic of Iowa, Cedar Rapids, Iowa
  - Holy Cross Hospital Holy Cross (2), Silver Spring, Maryland
  - Southeast Nebraska Oncology, Lincoln, Nebraska
  - Comprehensive Cancer Centers of Nevada CCC of Nevada (1), Las Vegas, Nevada
  - Duke University Medical Center Seeley G. Mudd Bldg., Durham, North Carolina
  - Wake Forest Baptist Health Health Sciences, Winston-Salem, North Carolina
  - Sanford Hematology Oncology, Fargo, North Dakota
  - Columbus Hematology and Oncology PA Columbus Hem and Onc (2), Columbus, Ohio
  - Andrew and Patel Associates, Camp Hill, Pennsylvania
  - Rhode Island Hospital Rhode Island Hosp. (2), Providence, Rhode Island
  - Sanford University of South Dakota Medical Center Sanford Clinical Research, Sioux Falls, South Dakota
  - Oncology Consultants Oncology Group, Houston, Texas
  - MD Anderson Cancer Center/University of Texas MD Anderson Cancer Center (3), Houston, Texas
  - Utah Cancer Specialists Utah Cancer Specialists, Salt Lake City, Utah
  - Swedish Cancer Institute Swedish Cancer Institute, Seattle, Washington
  - Aurora Research Institute, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ceritinib 750 mg
Started | 47
Completed | 0
Not Completed | 47
Not completed — Adverse Event | 9
Not completed — Death | 2
Not completed — Disease progression | 32
Not completed — Protocol Violation | 1
Not completed — Physician Decision | 1
Not completed — Study terminated by sponsor | 2

BASELINE CHARACTERISTICS:
Arm/Group | Ceritinib 750 mg
Number analyzed (Participants) | 47
Age, Customized [Count of Participants; unit: Participants]
  <65 | 27
  ≥65 - < 75 | 15
  ≥75 | 5
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female Able to bear children | 2
  Female Premenarche | 0
  Female Postmenopausal | 14
  Female Sterile of child bearing age | 6
  Male | 25
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 38
  Black | 2
  Asian | 3
  Native American | 1
  Other | 3
Participants with primary tumor type (sponsor adjudicated) [Count of Participants; unit: Participants] — Number of participants with primary type of tumor
  Participants
    Ampullary adenocarcinoma | 1
    Appendix | 1
    Breast | 2
    Central nervous system | 1
    Cervix | 1
    Colorectal cancer | 10
    Gastroesophageal junction | 1
    Head and neck squamous cell carcinoma | 1
    Liver | 1
    Lung non-small cell adenocarcinoma | 7
    Lymphoma | 1
    Neuroendocrine | 1
    Ovarian | 5
    Pancreas | 1
    Prostate | 1
    Sarcoma | 7
    Skin non-melanoma | 1
    Uterus | 2
    Uveal Melanoma | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Overall Response Rate (ORR) and Clinical Benefit Rate (CBR) Utilizing RECIST 1.1 at Approximately 16 Weeks
Description: Solid tumors were assessed using RECIST 1.1 criteria and included responses of complete response (CR) or partial response (PR) or stable disease (SD). For hematologic tumors, other hematological response criteria applied. CR=disappearance of all target lesions. Pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10mm. PR=at least 30% decrease in sum of diameters of target lesions from baseline sum diameters. SD=neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest sum diameters while on study. Progressive disease (PD)=at least a 20% increase in sum of diameter of measured target lesions from smallest sum of diameter of all target lesions recorded at or after baseline (sum must also demonstrate an absolute increase of at least 5mm). One or more new lesions was considered PD. Overall response rate (ORR) = (CR + PR). Clinical benefit rate = (CR + PR + SD)
Time Frame: Baseline up to approximately 16 weeks
Population: ORR and CBR was reported for all patients and for a subgroup of patients with colorectal cancer
Measure: Number (95% Confidence Interval); unit: percentage of paarticipants
Arm/Group | Ceritinib 750 mg
Number analyzed (Participants) | 47
percentage of paarticipants
  ORR (CR + PR) for all patients | 6.4 [1.3 to 17.5]
  CBR (CR + PR + SD) for all patients | 19.1 [9.1 to 33.3]
  ORR (CR + PR) for colorectal cancer patients: number analyzed (Participants) | 10
  ORR (CR + PR) for colorectal cancer patients | 0.0 [0.0 to 30.8]
  CBR (CR + PR + SD) for colorectal cancer: number analyzed (Participants) | 10
  CBR (CR + PR + SD) for colorectal cancer | 10.0 [0.3 to 44.5]

2. Primary Outcome: Number of Participants With Tumor Responses Utilizing RECIST 1.1 at Approximately 16 Weeks
Description: For patients with solid tumors the assessment criteria was RECIST 1.1 and included responses of complete response (CR) or partial response (PR) or stable disease (SD). For hematologic tumors, other hematological response criteria applied. CR=disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10mm. PR=at least a 30% decrease in sum of diameters of target lesions, taking as reference the baseline sum diameters. SD=neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest sum diameters while on study. Progressive disease (PD)=at least a 20% increase in sum of diameter of all measured target lesions, taking as reference the smallest sum of diameter of all target lesions recorded at or after baseline (sum must also demonstrate an absolute increase of at least 5mm). One or more new lesions was also considered progression.
Time Frame: Baseline up to approximately 16 weeks
Population: tumor response was reported for all patients and for a subgroup of patients with colorectal cancer
Measure: Count of Participants; unit: Participants
Arm/Group | Ceritinib 750 mg
Number analyzed (Participants) | 47
Participants
  Complete response - all patients | 0
  Partial response - all patients | 3
  Stable disease- all patients | 6
  Progressive disease - all patients | 32
  Non-evaluable - all patients | 6
  Stable disease - Colorectal cancer patients: number analyzed (Participants) | 10
  Stable disease - Colorectal cancer patients | 1
  PD - Colorectal cancer patients: number analyzed (Participants) | 10
  PD - Colorectal cancer patients | 8
  Non-evaluable - Colorectal cancer patients: number analyzed (Participants) | 10
  Non-evaluable - Colorectal cancer patients | 1

3. Secondary Outcome: Progression-Free Survival (PFS)
Description: Progression-free survival (PFS) was the time from the date of start of study drug to the date of event defined as the first documented progression or death due to any cause within 30 days of the last dose. If a patient has not had an event, progression-free survival was censored at the date of last adequate tumor assessment.
Time Frame: Baseline up to approximately 27 months
Population: reported for all patients and for a subgroup of patients with colorectal cancer
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ceritinib 750 mg
Number analyzed (Participants) | 47
months
  All patients: number analyzed (Participants) | 36
  All patients | 1.8 [1.5 to 1.9]
  Colorectal cancer patients: number analyzed (Participants) | 9
  Colorectal cancer patients | 1.8 [1.0 to 1.9]

4. Secondary Outcome: Percentage of Participants With Progression-Free Survival (PFS) - Kaplan-Meier Estimates
Description: as for outcome 3
Time Frame: Basleline up to approximately 27 months
Population: reported for all patients and for a subgroup of patients with colorectal cancer
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ceritinib 750 mg
Number analyzed (Participants) | 47
Percentage of participants
  1 Month | 81.0 [65.5 to 90.0]
  2 Month | 34.8 [20.8 to 49.2]
  3 Month | 34.8 [20.8 to 49.2]
  4 Month | 24.1 [12.3 to 38.2]
  5 Month | 21.4 [10.3 to 35.2]
  6 Month | 15.3 [6.0 to 28.6]
  9 Month | 11.5 [3.5 to 24.8]
  12 Month | 7.7 [1.6 to 20.5]
  18 Month | 7.7 [1.6 to 20.5]
  24 Month | 7.7 [1.6 to 20.5]
  30 Month | 7.7 [1.6 to 20.5]
  1 Month Colorectal cancer patients: number analyzed (Participants) | 10
  1 Month Colorectal cancer patients | 90.0 [47.3 to 98.5]
  2 Month Colorectal cancer patients: number analyzed (Participants) | 10
  2 Month Colorectal cancer patients | 12.5 [0.7 to 41.8]
  3 Month Colorectal cancer patients: number analyzed (Participants) | 10
  3 Month Colorectal cancer patients | 12.5 [0.7 to 41.8]
  4 Mongth Colorectal cancer patients: number analyzed (Participants) | 10
  4 Mongth Colorectal cancer patients | 12.5 [0.7 to 41.8]
  5 Month Colorectal cancer patients: number analyzed (Participants) | 10
  5 Month Colorectal cancer patients | 12.5 [0.7 to 41.8]
  6 Month Colorectal cancer patients: number analyzed (Participants) | 10
  6 Month Colorectal cancer patients | 12.5 [0.7 to 41.8]
  9 Month Colorectal cancer patients: number analyzed (Participants) | 10
  9 Month Colorectal cancer patients | 12.5 [0.7 to 41.8]

5. Secondary Outcome: Overall Survival (OS) - Number of Participant Deaths
Description: Overall survival (OS) is defined as the time from the date of first dose to the date of death due to any cause
Time Frame: Baseline up to approximately 27 months
Measure: Count of Participants; unit: Participants
Arm/Group | Ceritinib 750 mg
Number analyzed (Participants) | 47
Participants
  Deaths due to study indication | 14
  Deaths due to study indication while on treatment | 5

6. Secondary Outcome: Duration of Response (DOR)
Description: Duration of response (DOR) is defined as time from the first documented response (CR or PR) to the date first documented disease progression or relapse or death due to any cause
Time Frame: baseline up to approximately 30 months
Population: only 2 patients met criteria for duration of response
Measure: Number; unit: days
Arm/Group | Ceritinib 750 mg
Number analyzed (Participants) | 47
days
  One Patient with PR: number analyzed (Participants) | 1
  One Patient with PR | 132
  Second Patient with PR: number analyzed (Participants) | 1
  Second Patient with PR | 113

7. Post Hoc Outcome: All Collected Deaths
Description: On treatment deaths were collected from FPFT up to 30 days after study drug discontinuation, for a maximum duration of 27 months (treatment duration ranged from 0.2 to 25.9 months). Deaths post treatment survival follow up were collected after the on treatment period, up to approximately 39 months.
Time Frame: approx. 26 months, approx. 39 months
Population: Clinical Database Population: All treated patients
Measure: Number; unit: Participants
Arm/Group | Ceritinib 750 mg
Number analyzed (Participants) | 47
Participants
  Total deaths | 14
  Deaths on treatment | 5

ADVERSE EVENTS:
Time Frame: Adverse events were collected from FPFT up to 30 days after study drug discontinuation, for a maximum duration of 27 months (treatment duration ranged from 0.2 to 26.9 months).
Description: AE: Any sign or symptom that occurs during the study treatment plus the 30 days post treatment
Arm/Group | Ceritinib 750 mg
All-Cause Mortality (participants affected / at risk) | 5/47
Serious Adverse Events (participants affected / at risk) | 16/47
Other Adverse Events (participants affected / at risk) | 46/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ceritinib 750 mg (N=47)
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 3
Ileus (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Small intestinal obstruction (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Fatigue (General disorders) | 1
Malaise (General disorders) | 1
Pyrexia (General disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 2
Jaundice cholestatic (Hepatobiliary disorders) | 1
Clostridium difficile infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 3
Fall (Injury, poisoning and procedural complications) | 1
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 2
Blood alkaline phosphatase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Tongue neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Aphasia (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ceritinib 750 mg (N=47)
Anaemia (Blood and lymphatic system disorders) | 7
Abdominal distension (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 12
Constipation (Gastrointestinal disorders) | 9
Diarrhoea (Gastrointestinal disorders) | 36
Dyspepsia (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 33
Vomiting (Gastrointestinal disorders) | 24
Fatigue (General disorders) | 24
Oedema peripheral (General disorders) | 3
Hyperbilirubinaemia (Hepatobiliary disorders) | 3
Oral candidiasis (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 4
Alanine aminotransferase increased (Investigations) | 15
Aspartate aminotransferase increased (Investigations) | 19
Blood alkaline phosphatase increased (Investigations) | 13
Blood creatine phosphokinase increased (Investigations) | 3
Blood creatinine increased (Investigations) | 14
Electrocardiogram QT prolonged (Investigations) | 4
Gamma-glutamyltransferase increased (Investigations) | 12
Weight decreased (Investigations) | 7
Decreased appetite (Metabolism and nutrition disorders) | 17
Dehydration (Metabolism and nutrition disorders) | 6
Hyperglycaemia (Metabolism and nutrition disorders) | 4
Hyperuricaemia (Metabolism and nutrition disorders) | 5
Hypokalaemia (Metabolism and nutrition disorders) | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 6
Hyponatraemia (Metabolism and nutrition disorders) | 5
Back pain (Musculoskeletal and connective tissue disorders) | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Headache (Nervous system disorders) | 4
Chromaturia (Renal and urinary disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 6
Hypotension (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-04-09): https://cdn.clinicaltrials.gov/large-docs/21/NCT02186821/SAP_000.pdf
  • Study Protocol (2016-01-06): https://cdn.clinicaltrials.gov/large-docs/21/NCT02186821/Prot_001.pdf